CLINICAL TRIAL: NCT04589377
Title: Mobile Mindfulness Training and Physics Learning
Brief Title: Mindfulness to Mitigate Psychological Threat and Improve Engagement and Learning in Introductory Physics Courses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: U.S. National Science Foundation (U.S. Federal Agency); James S McDonnell Foundation (Other)
Responsible Party: Principal Investigator, Brian Galla, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY19050258 Part 1
Record Dates: First submitted 2020-10-08; First posted 2020-10-19 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Stress
Keywords: psychological threat; motivation; engagement; physics education; mindfulness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Training (Experimental): Participants receive 20 minutes of mindfulness training per day for five continuous days (Monday through Friday). Training is delivered remotely to participants' computers and smartphones.
  Interventions: Behavioral: Mindfulness Training
- No-Training (No Intervention): Participants do not receive training. On Monday and Friday, they listen to a 20 minute audiobook to match for time.

INTERVENTIONS:
Behavioral: Mindfulness Training — Training is focused on learning the principle of RAIN (recognize, accept, investigate, non-identify) in the context of physics learning.
  Arms: Mindfulness Training

SUMMARY:
This project involves testing a brief mindfulness training program to reduce students' psychological threat and support motivation, engagement, and learning in introductory undergraduate physics courses. The investigators predict that, compared to a control condition, mindfulness training will reduce psychological threat and increase motivation, engagement, and learning in physics.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* current University of Pittsburgh student
* fluent in written and spoken English
* enrolled in introductory physics
* self-reported psychological threat in physics

Exclusion Criteria:

* under 18 years of age
* not a current University of Pittsburgh student
* not fluent in written and spoken English
* not enrolled in introductory physics
* does not meet self-report psychological threat in physics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Mean differences in Psychological Threat measured via Ecological Momentary Assessment | Up to 3 days post-random assignment
  Perceived physics demands and physics coping resources, measured using self-report items with Likert scale from 1 to 6. Psychological threat is calculated by subtracting average of physics demands from average of physics resources. Psychological threat ranges from -5 to 5, with scores above zero indicating psychological threat and scores of 0 or lower indicating psychological challenge.
Mean differences in Physics Motivation assessed via Ecological Momentary Assessment | Up to 3 days post-random assignment
  State motivation to do physics work, measured using self-report items with Likert scale from 1 to 4. Physics motivation is calculated as an average of all items. Physics motivation ranges from 1 to 4, with higher scores indicating greater motivation to do physics work.
Mean change in Psychological Threat measured via Self-Report | Up to three months post-intervention
  Perceived physics demands and physics coping resources, measured using self-report items with Likert scale from 1 to 6. Psychological threat is calculated by subtracting average of physics demands from average of physics resources. Psychological threat ranges from -5 to 5, with scores above zero indicating psychological threat and scores of 0 or lower indicating psychological challenge.
Mean change in Physics Interest measured via Self-Report | Up to three months post-intervention
  The degree by which student's want to know or learn about physics, measured using self-report items with Likert scale from 1 to 4. Physics interest is calculated as an average of all items. Physics interest ranges from 1 to 4, with higher scores indicating greater interest in learning about physics.
Mean change in Physics Self-Efficacy measured via Self-Report | Up to three months post-intervention
  Beliefs about the ability to perform well in physics, measured using self-report items with Likert scale from 1 to 4. Physics self-efficacy is calculated as an average of all items. Physics self-efficacy ranges from 1 to 4, with higher scores indicated greater self-efficacy to perform well in physics.
Mean change in Physics Value measured via Self-Report | Up to three months post-intervention
  Perceived value of learning physics, measured using self-report items with Likert scale from 1 to 6. Physics value is calculated as an average of all items. Physics value ranges from 1 to 6, with higher scores indicating greater perceived value of physics learning.
Mean change in Physics Identity measured via Self-Report | Up to three months post-intervention
  The degree by which students identify their self-concept with physics, measured using self-report items with Likert scale from 1 to 6. Physics identity is calculated as an average of all items. Physics identity ranges from 1 to 6, with higher scores indicating greater self-identification with physics.
Mean change in Physics Belonging measured via Self-Report | Up to three months post-intervention
  Student's sense of belonging in their physics course, measured using self-report items with Likert scale from 1 to 5. Physics belonging is calculated as an average of all items. Physics belonging ranges from 1 to 5, with higher scores indicating greater sense of belonging in physics.
Mean change in Physics Achievement Goals measured via Self-Report | Up to three months post-intervention
  Goals related to mastery approach, performance approach, or performance avoidance, measured using self-report items with Likert scale from 1 to 6. Each subscale is calculated as an average of all of the items for each subscale. Physics achievement goals range from 1 to 6, with higher scores indicating greater mastery approach, performance approach, or performance avoidance goals.
Mean change in Physics Growth Mindset measured via Self-Report | Up to three months post-intervention
  Beliefs that intelligence and abilities for physics can be developed through dedication and hard work, measured using self-report items with Likert scale from 1 to 6. Growth mindset is calculated as an average of all items. Growth mindset ranges from 1 to 6, with higher scores indicating greater growth mindsets and lower scores indicating greater fixed mindsets.

SECONDARY OUTCOMES:
Mean differences in Meaning Making and Positive Reappraisal assessed via Ecological Momentary Assessment | Up to 3 days post-random assignment
  Positive Construals and appraisals of a difficult experience in physics, measured using self-report items with Likert scale from 1 to 5. Positive construals and appraisals are calculated as an average of all items. Positive construals and appraisals ranges from 1 to 5, with higher scores indicating greater positive reappraisal of a difficult experience in physics.
Mean differences in Affect assessed via Ecological Momentary Assessment | Up to 3 days post-random assignment
  Positive and negative affect, measured using self-report items with Likert scale from 1 to 5. Positive and negative affect are calculated as an average of all items from each subscale. Positive and negative affect ranges from 1 to 5, with higher scores indicating greater positive or negative affect, respectively.
Mean differences in Mindfulness assessed via Ecological Momentary Assessment | Up to 3 days post-random assignment
  State mindful attention and awareness, measured using self-report items with Likert scale from 0 to 6. State mindfulness is calculated as an average of all items. State mindfulness ranges from 0 to 6, with higher scores indicating greater state mindful attention and awareness.
Mean differences in Equanimity assessed via Ecological Momentary Assessment | Up to 3 days post-random assignment
  State balanced mental attitude, measured using self-report items with Likert scale from 1 to 5. State equanimity is calculated as an average of all items. State equanimity ranges from 1 to 5, with higher scores indicating a greater balanced mental attitude.
Mean change in Meaning Making and Positive Reappraisal assessed via Self-Report | Up to three months post-intervention
  Positive construals and appraisals of a difficult experience in physics, measured using self-report items with Likert scale from 1 to 5. Positive construals and appraisals are calculated as an average of all items. Positive construals and appraisals ranges from 1 to 5, with higher scores indicating greater positive reappraisal of a difficult experience in physics.
Mean change in Physics Engagement assessed via Self-Report | Up to three months post-intervention
  Physics effort, cognitive strategies, metacognitive strategies, & help-seeking, with each subscale measured using self-report items with Likert scale from 1 to 6. Each subscale is calculated as an average of all of the items for each subscale, with higher scores indicating greater effort, use of cognitive strategies, metacognitive strategies, and greater help-seeking behavior.
Mean change in Physics Anxiety assessed via Self-Report | Up to three months post-intervention
  Anxiety about doing physics work, measured using self-report items with Likert scale from 1 to 5. Physics anxiety is calculated as an average of all items. Physics anxiety ranges from 1 to 5, with higher scores indicating greater physics anxiety.
Mean change in Physics performance on the assessment | Change from baseline to posttest
  Physics problem solving tasks that range in difficulty covering content from introductory physics. Each item is scored for accuracy. Multiple choice and forced choice items scored as correct or incorrect. Open-ended and explanation items are scored on a rubric. Scores are averaged across the items with higher scores indicating better physics performance.
Mean differences in Performance on the Preparation for Future Learning Task | Posttest
  Physics problem solving tasks that include new learning resources (e.g., a worked example) and a transfer task. Each item is scored for accuracy. Open-ended and explanation items are scored on a rubric. Scores are summed across items with higher scores indicating better physics learning.
Mean change of judgments of confidence, anxiety, and difficulty during physics assessment via Self-Report | Change from baseline to posttest
  Judgments of anxiety, confidence, and difficulty during physics problem solving, with each subscale measured using self-report items with Likert scale from 1 to 6. Each subscale is calculated as an average of all of the items, with higher scores indicating greater confidence, anxiety, and difficulty respectively.

OTHER OUTCOMES:
Mean differences in Performance in Physics Class | End of semester, approximately 12 weeks
  End-of-course grades measured via school records on a scale from 0-4. Higher grades indicate higher classroom performance.
Mean differences in Retention in Physics Classes | End of following semester, approximately 7 months
  Enrollment in second semester of introductory physics course sequence measured via official school records. Scored dichotomously, 1 for enrolling in second semester physics and 0 for not.
Mean change in Physics Failure Mindset assessed via Self-Report | Up to three months post-intervention
  Perceptions of failure ranging from failure-is-enhancing to failure-is-debilitating, measured using self-report items with Likert scale from 1 to 5. Physics failure mindset is calculated as an average of all items. Physics failure mindset ranges from 1 to 6, with higher scores indicating a greater failure-is-debilitating mindset.
Mean change in Physics Epistemological Beliefs assessed via Self-Report | Up to three months post-intervention
  Beliefs about the nature of physics, measured using self-report items with Likert scale from 1 to 6. Physics beliefs is calculated as an average of all items. Physics beliefs ranges from 1 to 6, with higher scores indicating greater implementation of instruction and learning tools.
Mean change in Physics Transfer assessed via Self-Report | Up to three months post-intervention
  General self-reported learning and transfer strategies, measured using self-report items with Likert scale from 1 to 6. Physics transfer is calculated as an average of all items. Physics transfer ranges from 1 to 6, with higher scores indicating greater use of learning and transfer strategies.
Mean change in Covid-19 Perception of Threat assessed via Self-Report | Up to three months post-intervention
  Perceptions of threat due to Covid-19 and its relation to school, measured using self-report items with Likert scale from 1 to 6. Covid-19 perception of threat is calculated as an average of all items. Covid-19 perception of threat ranges from 1 to 6, with higher scores indicating greater perceived threat due to Covid-19.
Mean change in Mindfulness assessed via Self-Report | Up to three months post-intervention
  Trait mindful attention and awareness, measured using self-report items with Likert scale from 1 to 5. Trait mindfulness is calculated as an average of all items. Trait mindfulness ranges from 1 to 5, with higher scores indicating greater mindful attention and awareness; will also be used as covariate or moderator Trait mindful attention and awareness, measured using self-report items with Likert scale from 1 to 5. Trait mindfulness is calculated as an average of all items. Trait mindfulness ranges from 1 to 5, with higher scores indicating greater mindful attention and awareness; will also be used as covariate or moderator
Mean change in Emotion Regulation assessed via Self-Report | Up to three months post-intervention
  Trait emotion regulation and dysregulation, measured using self-report items with Likert scale from 1 to 5. Trait emotion regulation is calculated as an average of all items. Trait emotion regulation ranges from 1 to 5, with higher scores indicating greater regulation of emotions and lower scores indicating a dysregulation of emotions; will also be used as covariate or moderator
Mean change in Trait Equanimity assessed via Self-Report | Up to three months post-intervention
  Trait balanced mental attitude, measured using self-report items with Likert scale from 1 to 5. Trait equanimity is calculated as an average of all items. Trait equanimity ranges from 1 to 5, with higher scores indicating a greater balanced mental attitude; will also be used as covariate or moderator

CONTACTS AND LOCATIONS:
Overall Officials: Brian Galla, PhD, Principal Investigator — University of Pittsburgh; Timothy Nokes-Malach, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data required to reproduce results reported in publications will be available to researchers.
Supporting Information: Analytic Code
Time Frame: Data and analytic code will be shared upon publication.
Access Criteria: Data and analytic code will be shared on Open Science Framework (or other online repository)